CLINICAL TRIAL: NCT02190214
Title: Thyroid Disorders in Malaysian: A Nationwide Multicentre Study
Brief Title: Thyroid Disorders in Malaysia: A Nationwide Multicentre Study
Acronym: MyEndo-Thyroid
Status: Completed | Type: Observational
Sponsor: International Islamic University Malaysia (Other)
Collaborators: Malaysian Endocrine and Metabolic Society (Other); National University of Malaysia (Other); University of Malaya (Other); IMU University, Malaysia (Other)
Responsible Party: Principal Investigator, Dr Mohamnmad Arif Shahar, Assist Prof, International Islamic University Malaysia
Other Study IDs: MyEndo-Thyroid
Record Dates: First submitted 2014-07-09; First posted 2014-07-15 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Hypothyroidism; Subclinical Hypothyroidism; Hyperthyroidism; Subclinical Hyperthyroidism; Graves Disease; Hashimoto's Thyroiditis; Iodine Deficiency; Genetic Susceptibility
Keywords: Hyperthyroidism; Hypothyroidism; Autoimmune thyroid disorders; Iodine deficiency; Genetic susceptibility
MeSH Terms: conditions — Hypothyroidism; Hyperthyroidism; Graves Disease; Hashimoto Disease; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood Serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This will be a population based study looking at the prevalence of thyroid disorders in Malaysia (including hypo- and hyperthyroidism, subclinical hypo- or hyperthyroidism) and its association with different ethnicity and iodine status. The study will also look at genetic susceptibility for autoimmune thyroid disorders in the Malaysian population

General hypotheses:

The prevalence of thyroid disorders in Malaysia is 10% for hypothyroidism and 2% for hyperthyroidism Hypo- and hyperthyroidism is associated with iodine status in our population There are different susceptibility gene for autoimmune thyroid disorder in different ethnicity in our population

DETAILED DESCRIPTION:
This will be a cross-sectional population based study involving Malaysian adults (aged 18 year old and above). Cluster sampling will be used to select respondents that will be representative of the Malaysian population. Selected respondent will be interviewed, anthropometric measurement taken, blood and urine sample taken.

Blood will be analyzed for thyroid function (thyroxine, triiodothyronine and thyroid stimulating hormone), autoantibodies (anti-thyroperoxidase and anti-thyroglobulin). Urine will be analyzed for urinary iodine.

Those diagnosed with autoimmune thyroid disorders with strong family history of thyroid disorders (multiplex multi-generation family involvement) will have their blood sent for whole exome sequencing and linkage analysis done to identify possible susceptible gene for autoimmune thyroid disorders

Respondents detected to have hypo- or hyper- and subclinical hypo- or hyperthyroidism will be referred to their nearest health centre for further evaluation and treatment appropriate for their condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged equal or more than 18 years old at the time of sampling
* Malaysian citizen

Exclusion Criteria:

* Respondents who did not give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult (aged equal or more than 18 years old ) Malaysian citizen living in Malaysia at the time of sampling
Sampling Method: Probability Sample
Enrollment: 2498 (Actual)
Dates: Start 2014-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal thyroid function | Day 0
  Overt or subclinical hypothyroidism Overt or subclinical hyperthyroidism

SECONDARY OUTCOMES:
Number of participants with positive thyroid autoantibodies | Day 0
  Anti-thyroglobulin Anti-thyroperoxidase
Number of participants with Iodine deficiency status | Day 0
  Urinary iodine level

OTHER OUTCOMES:
Number of participants with genetic susceptibility to autoimmune thyroid disorders | Day 0
  whole exome sequencing and linkage analysis in families with autoimmune thyroid disorders (multiplex multi-generation involvement)

CONTACTS AND LOCATIONS:
Overall Officials: Nor Azmi Kamaruddin, MBBS, MMed, Principal Investigator — National University of Malaysia; Norlela Sukor, MMed, Phd, Principal Investigator — National University of Malaysia; Norhanita Othman, Principal Investigator — National University of Malaysia; Johari Ali, Principal Investigator — University of Malaya; Shirenee Vethakkan, Principal Investigator — University of Malaya; Siew Kim Kwa, Principal Investigator — IMU University, Malaysia; Kuck Meng Chong, MD, Principal Investigator — Malaysian Endocrine and Metabolic Society; Lecthuman Ramanathan, Principal Investigator — Malaysian Endocrine and Metabolic Society; Hussein Zanariah, Principal Investigator — Malaysian Endocrine and Metabolic Society; Nurain Mohd Noor, Principal Investigator — Malaysian Endocrine and Metabolic Society; Norhaliza Mohd Ali, Principal Investigator — Malaysian Endocrine and Metabolic Society; Norhayati Yahya, Principal Investigator — Malaysian Endocrine and Metabolic Society; Nor Azizah Aziz, Principal Investigator — Malaysian Endocrine and Metabolic Society